CLINICAL TRIAL: NCT03466151
Title: A Randomized Controlled Trial to Evaluate the Safety and Efficacy of the Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System in Comparison With the Medtronic Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System in the Treatment of Subjects Eligible for Percutaneous Transluminal Coronary Angioplasty (PTCA) in China
Brief Title: RESOLUTE ONYX China RCT Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT16061RES005
Record Dates: First submitted 2018-03-01; First posted 2018-03-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Heart Disease; Stenotic Coronary Lesion; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease
Keywords: Major Adverse Cardiac Events (MACE); Myocardial Infarction (MI); Late Lumen Loss (LLL); Target Lesion Revascularization (TLR); Target Vessel Revascularization (TVR); Target Vessel Failure (TVF); Target Lesion Failure (TLF); Stent Thrombosis (ST); The Randomized Controlled Trial; PERCUTANEOUS CORONARY INTERVENTION (PCI)
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System (Experimental): Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System
  Interventions: Device: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System
- Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System (Active Comparator): Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System
  Interventions: Device: Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System — Treatment of subjects eligible for percutaneous transluminal coronary angioplasty (PTCA) as per study requirements
  Arms: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System
Device: Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System — Treatment of subjects eligible for percutaneous transluminal coronary angioplasty (PTCA) as per study requirements
  Arms: Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System

SUMMARY:
It is a randomized controlled trial to evaluate the safety and efficacy of the Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System in comparison with the Medtronic Resolute Integrity™ Zotarolimus-Eluting coronary stent system in the treatment of subjects eligible for percutaneous transluminal coronary angioplasty (PTCA) in China.

DETAILED DESCRIPTION:
This study is a pre-Market, prospective, multi-center, open-label, randomized controlled trial. Subjects will be 1:1 randomized and followed through 5 Years (screen, implant procedure(including post-procedure assessment),30-Day, 6 Months, 9 Months (primary endpoint_LLL), and annual assessments from 1-5 years).

ELIGIBILITY:
Key Inclusion Criteria:

* The subject is an acceptable candidate for treatment with a drug-eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, the IB of Resolute Onyx stent, and the IFU of Resolute Integrity stent
* The subject requires treatment of up to 3 target lesions in up to 2 separate target vessels [2 target lesions in 1 vessel (including its side branches) and 1 target lesion in a separate vessel(including its side branches)] amenable to treatment with stents with diameter from 2.25 mm to 4.0 mm

Key Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, P2Y12 inhibitors, mTOR inhibiting drugs such as zotarolimus, Biolimus A9 (or its derivatives), cobalt, nickel, platinum, iridium, chromium, molybdenum, polymer coatings (e.g. BioLinx) or a sensitivity to contrast media, which cannot be adequately pre-medicated
* PCI of the target vessel within 9 months prior to the procedure
* Active bleeding
* Subjects with a life expectancy of less than 12 months
* Participation in another clinical study
* Pregnant, or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
In-stent Late lumen loss measured by quantitative coronary angiography (QCA) | 9 months
  Late lumen loss measured by quantitative coronary angiography (QCA)

SECONDARY OUTCOMES:
Device Success | at the end of the index procedure or during hospital stay: estimated 7 days
  Definition 1: The attainment of <50% residual stenosis of the target lesion using only the assigned device.
  Definition 2: The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using the assigned device only. These measurements will be made by the independent angiographic core laboratory.
Lesion Success | at the end of the index procedure or during hospital stay: estimated 7 days
  Definition 1: The attainment of <50% residual stenosis of the target lesion using any percutaneous method.
  Definition 2: The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using the assigned device only. These measurements will be made by the independent angiographic core laboratory.
Procedure Success | at the end of the index procedure or during hospital stay: estimated 7 days
  Definition 1: The attainment of <50% residual stenosis of the target lesion and no in-hospital MACE.
  Definition 2: The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using the assigned device only. These measurements will be made by the independent angiographic core laboratory.
Major Adverse Cardiac Events (MACE) | 30 day, 6 months, 9 months, 1 year, 2 years,3 years, 4 years, 5 years
  Defined as composite of death, myocardial infarction (Q wave and non-Q wave), emergent coronary bypass surgery, or clinically-driven repeat target lesion revascularization by percutaneous or surgical methods
Death (Cardiac and Non-cardiac) | 30 day, 6 months, 9 months, 1 year, 2 years,3 years, 4 years, 5 years
  All deaths
Myocardial infarction (all MI, and Target Vessel Myocardial Infarction (TVMI)) | 30 day, 6 months, 9 months, 1 year, 2 years,3 years, 4 years, 5 years
  All myocardial infarction data will be reported per Medtronic historical protocol definitions.
All revascularizations | 30 day, 6 months, 9 months, 1 year, 2 years,3 years, 4 years, 5 years
  Target Legion Revascularization (TLR), Target Vessel Revascularization (TVR) and Non-TVR
Target Vessel Failure (TVF) | 30 day, 6 months, 9 months, 1 year, 2 years,3 years, 4 years, 5 years
  TVF
Target Lesion Failure (TLF) | 30 day, 6 months, 9 months, 1 year, 2 years,3 years, 4 years, 5 years
  TLF
Stent Thrombosis (ST) | 30 day, 6 months, 9 months, 1 year, 2 years,3 years, 4 years, 5 years
  ST
In-stent and in-segment percent diameter stenosis (%DS) | 9 months
  Angiographic measures: In-stent and in-segment percent diameter stenosis (%DS)
In-stent and in-segment binary restenosis rate | 9 months
  Angiographic measures:In-stent and in-segment binary restenosis rate
In-stent and in-segment minimal luminal diameter (MLD) | 9 months
  Angiographic measures:In-stent and in-segment minimal luminal diameter (MLD)
In-segment late luminal loss | 9 months
  Angiographic measures: In-segment late luminal loss

CONTACTS AND LOCATIONS:
Overall Officials: Yongjian Wu, MD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Science
Locations (2):
- China (2):
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Fuwai Hospital, Chinese Academy of Medical Science, Beijing

DOCUMENTS (2):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT03466151/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT03466151/SAP_001.pdf